CLINICAL TRIAL: NCT04204005
Title: Probiotics-addicted Low-protein Diet for Microbiota Modulation in Patients With Advanced Chronic Kidney Disease (ProLowCKD): a Protocol of Placebo-controlled Randomized Trial
Brief Title: Probiotics and Low Protein Diet in Advanced Chronic Kidney Disease
Acronym: ProLowCKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Probiotical S.p.A. (Industry)
Collaborators: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 215/CE n.CE 30\17
Record Dates: First submitted 2019-11-29; First posted 2019-12-18 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2019-12

CONDITIONS: Renal Failure Chronic
Keywords: Low protein diet; Chronic kidney disease; Gut microbiota; Microbial uremic toxins; Probiotic bacteria; Intestinal dysbiosis
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: Single-centre, double-blind, placebo-controlled, randomised study.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Active Comparator): Composition: 5x109 of Bifidobacterium longum (mix DLBL), 1x109 Lactobacillus reuteri LRE02 (DSM 23878) and maltodextrin (total 2 grams)
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Composition: maltodextrin (2 grams)
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Active composition: 5x109 of Bifidobacterium longum (mix DLBL), 1x 109 Lactobacillus reuteri LRE02 (DSM 23878) and maltodextrin (total 2 grams). The probiotic species employed were granted the Qualified Presumption of Safety (QPS) status by the European Food Safety Authority (EFSA) in 2007. Two envelopes per day and one envelope per day will be recommended for one and two months, respectively.
  Placebo composition: maltodextrin (2 grams). Two envelopes per day and one envelope per day will be recommended for one and two months, respectively.

SUMMARY:
Here the investigators will perform a double-blinded randomized placebo-controlled clinical trial to evaluate the synergic effect of low protein diet and prebiotics in reducing the microbial inflammatory uremic toxins.

DETAILED DESCRIPTION:
ProLowCKD is a single-centre, double-blind, placebo-controlled, randomised study. At enrolment (T0) participants were prescribed a LPD in addition to their ongoing pharmacological therapy and according to their comorbidities; after 2 months (T2) they were randomized in accordance to a 1:1 ratio to receive probiotics or placebo for other 3 months (T5) in addition to the continuation of LPD. Enrolled subjects are invited to assume two doses of probiotic/placebo for 1 month and 1 dose for 2 months.

Randomization is 1:1 to receive odd- or even envelopes, according to the odd- or even registration number at enrolment.

Neither the clinician nor the patient knows the content of the odd- and even envelopes.

The evaluations will be performed according to the following schedule: at T0 nephrological evaluation and biochemical analysis, dietary counselling, illustration of protocol and signing of the informed consent, administration of the SF36 questionnaire, body composition evaluation by bioimpedentiometry. At T0, T2, T5: blood biochemical parameters: haemoglobin, urea, creatinine, mean urea and creatinine clearance, CKD and MDRD calculation, sodium, potassium, uric acid, calcium, phosphate, PTH, acid-base balance, CRP, albumin, PC, IS, Lp-PLA2, LPS; 24h-urine biochemical parameters: urea, creatinine, sodium, proteins; microbial stools analysis; clinical nephrological and dietitian evaluation.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80 years
* GFR < 20 ml/min/sqm
* afferent to the outpatient clinic in the Nephrology and Dialysis Unit (Azienda Ospedaliero Universitaria Maggiore della Carità)

Drop out or Exclusion Criteria:

* subject refusing to sign the informed consent
* administration of prolonged antibacterial therapy
* dialysis initiation
* death

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the microbial gut populations | 5 months
  * Change from baseline of the concentration of proteolytic microbial groups (number of cells/gram of faeces);
  * Change from baseline of the concentration of saccharolytic microbial groups (number of cells/gram of faeces)
Change from baseline of the microbial inflammatory uremic toxins | 5 months
  Change from baseline of the serum concentration of PC (mcMOL) and IS (mcMOL), as markers of dysbiotic microbiota
Change from baseline of the markers of cardiovascular diseases | 5 months
  Change from baseline of the serum concentration of Lp-PLA2 (nmol/ml/min)
Change from baseline of the markers of intestinal barrier permeability | 5 months
  Change from baseline of the serum concentration of LPS (EU/ml)

SECONDARY OUTCOMES:
Evaluation of the renal function | 5 months
  Change from baseline of ΔGFR (mL/min/m2 of body surface)
Measurement of the urine protein excretion | 5 months
  Change from baseline of 24-hour protein urine excretion (mg/24 hours)
Evaluation of the anemia | 5 months
  Change from baseline of haemoglobin (g/dL)
Evaluation of the serum acid-base equilibrium | 5 months
  Change from baseline of bicarbonatemia (mEq/l)
Quantification of serum inflammatory markers | 5 months
  Change from baseline of the serum concentration of C-reactive protein (CRP) (mg/dL)
Evaluation of the body composition | 5 months
  Change from baseline of fat-free body mass (kg), fat-body mass (kg), Hand Grip strength (kg), total body water (kg)
Measurement of vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health (Quality of Life) | 5 months
  Change from baseline of SF36 questionnaire score. The SF36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability.

CONTACTS AND LOCATIONS:
Overall Officials: Andreana De Mauri, Principal Investigator — Azienda Ospedaliero Universitaria Maggiore della Carità
Locations (1):
- Nephrology and Dialysis Unit, Azienda Ospedaliero Universitaria Maggiore della Carità, Novara, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marchesi JR, Adams DH, Fava F, Hermes GD, Hirschfield GM, Hold G, Quraishi MN, Kinross J, Smidt H, Tuohy KM, Thomas LV, Zoetendal EG, Hart A. The gut microbiota and host health: a new clinical frontier. Gut. 2016 Feb;65(2):330-9. doi: 10.1136/gutjnl-2015-309990. Epub 2015 Sep 2. PMID 26338727
- [Background] Ramezani A, Massy ZA, Meijers B, Evenepoel P, Vanholder R, Raj DS. Role of the Gut Microbiome in Uremia: A Potential Therapeutic Target. Am J Kidney Dis. 2016 Mar;67(3):483-98. doi: 10.1053/j.ajkd.2015.09.027. Epub 2015 Nov 15. PMID 26590448
- [Background] Mafra D, Fouque D. Gut microbiota and inflammation in chronic kidney disease patients. Clin Kidney J. 2015 Jun;8(3):332-4. doi: 10.1093/ckj/sfv026. Epub 2015 May 6. PMID 26034597
- [Background] Mafra D, Lobo JC, Barros AF, Koppe L, Vaziri ND, Fouque D. Role of altered intestinal microbiota in systemic inflammation and cardiovascular disease in chronic kidney disease. Future Microbiol. 2014;9(3):399-410. doi: 10.2217/fmb.13.165. PMID 24762311
- [Background] Rossi M, Klein K, Johnson DW, Campbell KL. Pre-, pro-, and synbiotics: do they have a role in reducing uremic toxins? A systematic review and meta-analysis. Int J Nephrol. 2012;2012:673631. doi: 10.1155/2012/673631. Epub 2012 Dec 19. PMID 23316359
- [Background] Vaziri ND. Effect of Synbiotic Therapy on Gut-Derived Uremic Toxins and the Intestinal Microbiome in Patients with CKD. Clin J Am Soc Nephrol. 2016 Feb 5;11(2):199-201. doi: 10.2215/CJN.13631215. Epub 2016 Jan 15. No abstract available. PMID 26772192
- [Derived] Cooper TE, Khalid R, Chan S, Craig JC, Hawley CM, Howell M, Johnson DW, Jaure A, Teixeira-Pinto A, Wong G. Synbiotics, prebiotics and probiotics for people with chronic kidney disease. Cochrane Database Syst Rev. 2023 Oct 23;10(10):CD013631. doi: 10.1002/14651858.CD013631.pub2. PMID 37870148